CLINICAL TRIAL: NCT03813966
Title: Self- and Parent/Guardian-Collection of Specimens for Rapid Influenza Nasal Swab Home Collection Kit (NSHC Kit) Study
Brief Title: Nasal Swab Home Collection Kit (NSHC Kit) Study
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Quidel Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 2018-1550; A532050 (Other: UW Madison); SMPH/FAMILY MEDICINE (Other: UW Madison)
Record Dates: First submitted 2019-01-15; First posted 2019-01-23 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-10

CONDITIONS: Influenza Viral Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Sofia Influenza A+B FIA — The Nasal Swab Home Collection Kit (NSHC Kit) provides the materials and training needed for you to safely collect a nasal swab at home. The sample can then be delivered to a designated test site for influenza testing.

SUMMARY:
The purpose of this study is to demonstrate that persons over the age of 13 years can obtain a self-collected nasal swab reliably and safely for subsequent use in the diagnosis of influenza. Similarly, the purpose is to demonstrate that parents or guardians can safely and effectively collect nasal swab specimens from children, ages 0 through 12 years, and others needing assistance in doing so, and that these parent/guardian-collected nasal swabs can also be used in the diagnosis of influenza. Clinical performance of the swabs will be based on the comparison of the performance of the nasal swab that is self- or parent/guardian-collected to one collected from the same specimen donor by a skilled clinical coordinator and used in CLIA (Clinical Laboratory Improvement Amendments)-waived, rapid diagnostic test called Sofia Influenza A+B FIA (fluorescence immunoassay analyzer).

ELIGIBILITY:
Inclusion Criteria:

* Fever
* Nasal Congestion
* Rhinorrhea
* Sore Throat
* Cough

Exclusion Criteria:

* Unable to read and understand or refusal to sign the appropriate informed consent/assent forms
* Refusal to complete the patient's demographic and medical history
* Treatment with anti-influenza antivirals within the previous 7 days
* Vaccinated by means of an influenza nasal spray/mist vaccine within the previous 7 days.

Min Age: 0 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: A maximum of 1,000 patients, representing the random ages of the patients presenting at the Urgent Care facilities, will be enrolled.
Sampling Method: Probability Sample
Enrollment: 1181 (Actual)
Dates: Start 2019-02-07 (Actual); Primary Completion 2020-03-04 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Diagnostic specificity of self-collected to technician collected nasal swab samples | 1 day (Participant); 17 weeks (Study length)
  Hypothesis tested is that self-collected nasal swab are as accurate as nasal swabs collected by a trained healthcare worker for the diagnosis of influenza by CLIA-waived, rapid diagnostic test called Quidel Sofia Influenza A+B Fluorescent Immunoassay. The investigators will specifically measure the specificity of self-collected specimens as compared to the clinical standard (trained healthcare worker collected specimen), estimating it using standard methods along with 95th% confidence intervals.
Diagnostic sensitivity of self-collected to technician collected nasal swab samples | 1 day (Participant); 17 weeks (Study length)
  Hypothesis tested is that self-collected nasal swab are as accurate as nasal swabs collected by a trained healthcare worker for the diagnosis of influenza by CLIA-waived, rapid diagnostic test called Quidel Sofia Influenza A+B Fluorescent Immunoassay. The investigators will specifically measure the sensitivity of self-collected specimens as compared to the clinical standard (trained healthcare worker collected specimen), estimating it using standard methods along with 95th% confidence intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Temte, MD PhD, Principal Investigator — University of Wisconsin, Madison
Locations (2):
- United States (2):
  - UWHealth Urgent Care Clinics, Madison, Wisconsin
  - UW Health Urgent Care Clinics, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No